CLINICAL TRIAL: NCT02884869
Title: Establishing a Definitive Airway: Comparison of Direct Laryngoscopy With Blind Intubation Via Intubating Laryngeal Mask Airway
Brief Title: Comparison of Direct Laryngoscopy With Blind Intubation Via Intubating Laryngeal Mask Airway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-006
Record Dates: First submitted 2016-08-16; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Blind intubation,; Laryngeal Mask Airway

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubating laryngeal Mask (Experimental): Intubating laryngeal Mask
  Interventions: Device: Intubating Laryngeal Mask
- Direct laryngoscopy (Active Comparator): Intubating laryngeal Mask
  Interventions: Device: Intubating Laryngeal Mask

INTERVENTIONS:
Device: Intubating Laryngeal Mask — Direct laryngoscopy

SUMMARY:
Control the airways by endotracheal intubation is an important part of treatment for a trauma casualty. The use of the Laryngeal Mask Airway for fast control of the airway is known for many years. The aim of this study is to examine the effectiveness of the Intubating Laryngeal Mask Airway to achieve a definitive airway by unskilled practitioners.

The hypothesis is that definitive airway obtaining with Intubating Laryngeal Mask Airway will be more success and faster compared to the standard way of direct laryngoscope.

DETAILED DESCRIPTION:
Control the airways and respiration are an important part of treatment for a trauma casualty. Tracheal intubation an action that allows the insertion of a tube through the vocal cords and fixation by the balloon inflation is a definitive airway. The use of the Laryngeal Mask Airway for fast control of the airway is known for many years. The Laryngeal Mask Airway and others similar devices are known as Supraglottic Airway Devices and are inserted blind in the oropharynx and allow a fast oxygenation and ventilation of the patients.The aim of this study is to examine the effectiveness of the Laryngeal Mask Airway to achieve a definitive airway by unskilled practitioners in anesthetized patients with the head in neutral position (trauma model)

The hypothesis is that definitive airway obtaining with Intubating Laryngeal Mask Airway will be more success and faster compared to the standard way of direct laryngoscope. If the hypothesis is proven, this research will be very important implications for the management of the airway describing pre-hospital and in particular military scenarios.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology class I and II

Exclusion Criteria:

* Difficult airway
* Cervical pathology
* Full stomach

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Time of blind intubation measure in second | 30 seconds
  Time of blind intubation in seconds

SECONDARY OUTCOMES:
Easy to perform intubation measure in numeric scale | 30 seconds
  Easy of intubation in numerical scale from 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Gaitini, M.D., Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Yes